CLINICAL TRIAL: NCT06669676
Title: Effect of Acupuncture on Postoperative Nausea and Vomiting in Lumbar Disc Herniation Surgeries
Brief Title: Effect of Acupuncture on Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Gökhan Erdem, Anesthesiology and Reanimation specialist doctor, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PONV
Record Dates: First submitted 2024-10-31; First posted 2024-11-01 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Anesthesia; Nausea and Vomiting, Postoperative
Keywords: acupuncture; postoperative nausea vomiting; apfel score
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture (Active Comparator): patients will be given acupuncture in addition to standard medical treatment to prevent ponv
  Interventions: Other: acupuncture
- No Acupuncture (Active Comparator): patients will be given acupuncture in addition to standard medical treatment to prevent ponv
  Interventions: Other: No acupuncture

INTERVENTIONS:
Other: acupuncture — patients will be given acupuncture in addition to standard medical treatment to prevent ponv
  Arms: Acupuncture
Other: No acupuncture — patients will be given standard medical treatment to prevent ponv
  Arms: No Acupuncture

SUMMARY:
In this study, the hypothesis that bilateral acupuncture needling at the Neiguan (PC6) point during the intraoperative period, in addition to the 0.15 mg/kg dose of ondansetron (5-HT3 antagonist) frequently used for postoperative nausea and vomiting (PONV) prophylaxis in patients undergoing lumbar disc herniation surgery, would reduce the incidence of PONV was investigated. PONV was defined as the presence of nausea and vomiting within 24 hours postoperatively.

DETAILED DESCRIPTION:
The study will include patients aged 18 years and over, with (American Society of Anesthesiologists) ASA physical status I to II, and scheduled for one or two-level lumbar disc herniation surgery under general anesthesia. Patient characteristics (age, gender, body mass index, etc.) and postoperative nausea and vomiting (PONV) risk factors such as history of PONV, motion sickness, and history of not smoking will be recorded. The primary outcome parameter will be the incidence of PONV within 24 hours postoperatively. The severity of nausea in patients who develop nausea in the postoperative period will be assessed using a Likert scale between 0 and 10. PONV will be defined as vomiting, significant nausea (numerical rating scale [NRS] ≥4), and/or need for rescue medication. Patients will be assessed for PONV at 0, 2, 4, 12, and 24 hours using a Likert scale. Emetic attacks, pain and severity of pain, nausea and severity of nausea, need for additional analgesics, and administration of antiemetic rescue medication will be assessed as secondary outcome parameters. The severity of pain and nausea in patients who develop postoperative pain will be assessed using an 11-point numerical rating scale, where '0' indicates the absence of symptoms and '10' indicates the maximum severity. PONV within the first two hours will be defined as 'early', and within 2-24 hours after awakening will be defined as 'late'. Nausea will be defined as the desire to vomit, and vomiting will be defined as the forceful expulsion of stomach contents.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and above
* ASA physical status I to II
* One or two level lumbar disc herniation surgery under general anesthesia

Exclusion Criteria:

* body mass index >35 kg/m²)
* history of drug use
* nausea and vomiting before surgery
* psychiatric disorders
* use of antipsychotic or antiemetic drugs
* severe heart disease
* central nervous system diseases
* vertebrobasilar artery insufficiency
* cytostatic therapy
* vestibular diseases
* renal and/or hepatic dysfunction
* presence of fistula, neuropathy and paralysis in the extremity to be treated
* patient's refusal to accept acupuncture
* pregnant patients
* presence of bleeding diathesis
* patients in a condition where cooperation cannot be established in the post-operative period (mental retardation etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-11-07 (Actual); Primary Completion 2025-02-15 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
PONV | 24 hours
  The primary outcome of the study was the incidence of postoperative nausea and/or vomiting

SECONDARY OUTCOMES:
Severity of nausea | 24 hours
  The degree of nausea was evaluated using the visual analogue scale (VAS), with 0 indicating no nausea or vomiting and 10 indicating the most severe form of unbearable nausea or vomiting. When the PONV score was greater than 4 or vomiting occurs
11 - point numerical rating scale (NRS) | 24 hours
  11-point numerical rating scale for pain (0='no pain' and 10='worst pain possible pain') were explained.
Rescue emetic requirement | 24 hours
  Number of additional emetic applications

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Ankara, Çankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No